CLINICAL TRIAL: NCT03960216
Title: Effects of Periodontal Therapy on Local and Systemic Markers of Inflammation in Patients With Metabolic Syndrome
Brief Title: Effects of Periodontal Therapy in Patients With Metabolic Syndrome
Acronym: MetS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12/206 CEIC Hospital Clínico
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Periodontitis; Metabolic Syndrome
MeSH Terms: conditions — Periodontitis; Metabolic Syndrome | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Periodontal Treatment (MPT) (Sham Comparator): Once the hopeless teeth have been extracted, randomized patients will receive a periodontal prophylaxis, in the form of supragingival removal of all deposits (plaque and calculus) with an ultrasonic scaler in two sessions, 1 week apart. During this week the patients will be prescribed local antiseptics (chlorhexidine rinse, 2x, 10 days) and, after the last session, placebo capsules (one every 24 h for three days).
  Interventions: Procedure: Supragingival Prophylaxis
- Intensive Periodontal Treatment (IPT) (Experimental): Once the hopeless teeth have been extracted, randomized patients will receive non-surgical periodontal therapy in the form of full-mouth scaling and root planing (SRP), in two sessions, 1 week apart, with the use of an ultrasonic scaler (Minipiezon Electromedical Systems EMS, Nyon, Switzerland) and hand instruments, under local anaesthesia. During this week the patients will be prescribed local antiseptics (chlorhexidine rinse, 2x, 10 days) and after the last session, systemic antibiotics (azithromycin 500 mgrs, every 24 h for three days).
  Interventions: Procedure: Scaling and root planning

INTERVENTIONS:
Procedure: Scaling and root planning — Patients received non-surgical periodontal therapy in the form of full-mouth scaling and root planing (SRP), in two sessions, 1 week apart, with the use of an ultrasonic scaler (Minipiezon Electromedical Systems EMS, Nyon, Switzerland) and hand instruments, under local anaesthesia.
  Arms: Intensive Periodontal Treatment (IPT)
Procedure: Supragingival Prophylaxis — Supragingival removal of all deposits (plaque and calculus) with an ultrasonic scaler in two sessions, 1 week apart.
  Arms: Minimal Periodontal Treatment (MPT)

SUMMARY:
A 6-month, parallel-arm, investigator-masked, randomized clinical trial was conducted in patients with MetS and severe periodontitis. Participants were randomly assigned to an Intensive Periodontal Treatment group (IPT; scaling and root planing and azithromycin capsules 500mg/24h/3days) or to a Minimal Periodontal Treatment group (MPT; professional plaque removal and placebo capsules). Blood and subgingival microbiological samples were collected at baseline, 3 and 6 months after therapy. The primary outcome was between-group difference in C-reactive protein (CRP). Secondary outcomes included HbA1c, lipids, α-1 antitrypsin, fibrinogen levels and subgingival microbiota assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Metabolic Syndrome according to the IDF definition
* at least 16 teeth
* at least eight sites with probing pocket depth (PPD) ≥ 6 mm and four sites with clinical attachment loss ≥ 5 mm, distributed in at least two different quadrants (Koromantzos et al. 2012).

Exclusion Criteria:

* They are not medically controlled for obesity and cardiovascular risk factors at the start of the study. For ethical reasons, patient inclusion must be delayed at least 3 months when begins a pharmacological treatment.
* They had history of kidney disease with Cr>1.2, CKD-EPI< 70 mil/min, or proteinuria > 300 mg/24 hours or 0.3 mg/grCr in isolated sample.
* They had history of chronic lung disease, or acute disease during the previous 3 months.
* They had history of stroke during the previous 3 months, myocardial infarction or revascularization during the previous 6 months, or recent angor pectoris history.
* They had history of known peripheral artery disease, or chronic heart failure.
* They had surgical treatment during the previous 3 months.
* They had any disease that conditions compliance along the study, such as alcoholism or psychiatric disorder.
* They had a history of systemic antibiotic usage over the previous 3 months.
* They had non-surgical periodontal treatment during the previous 6 months; or surgical periodontal treatment over the previous 12 months.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2013-05-30 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Change in C-reactive protein | Baseline, 3 months and 6 months
  Main outcome variable is the change in concentration of C-reactive protein between baseline and 6 months

SECONDARY OUTCOMES:
Change in Probing Pocket Depth | Baseline, 3 months and 6 months
  Examination of probing pocket depth will be determined with a periodontal probe and expressed in mm
Change in Clinical Attachment Level | Baseline, 3 months and 6 months
  Examination of clinical attachment level will be determined with a periodontal probe and expressed in mm
Change in Plaque Index | Baseline, 3 months and 6 months
  Examination of plaque index
Change in Bleeding on Probing | Baseline, 3 months and 6 months
  Examination of bleeding on probing
Change in the presence of selected periodontal pathogens | Baseline, 3 months and 6 months
  Selected periodontal pathogens: Aggregatibacter actinomycetemcomitans, Tannerella forsythia, P.gingivalis, Prevotella intermedia/nigrescens, Parvimonas micra, Campylobacter rectus and Fusobacterium nucleatum
Change in the total counts of selected periodontal pathogens | Baseline, 3 months and 6 months
  By means of anaerobic culture. Selected periodontal pathogens: Aggregatibacter actinomycetemcomitans, Tannerella forsythia, P.gingivalis, Prevotella intermedia/nigrescens, Parvimonas micra, Campylobacter rectus and Fusobacterium nucleatum
Change in the proportions of selected periodontal pathogens | Baseline, 3 months and 6 months
  Selected periodontal pathogens: Aggregatibacter actinomycetemcomitans, Tannerella forsythia, P.gingivalis, Prevotella intermedia/nigrescens, Parvimonas micra, Campylobacter rectus and Fusobacterium nucleatum
Change in the concentration of Inflammatory mediators (IL-1β, IL-6, IL-8 and TNF-α) in plasma and gingival crevicular fluid | Baseline, 3 months and 6 months
  The inflammatory mediators will be determined by Luminex
Change in the % of Glycated haemoglobin | Baseline, 3 months and 6 months
  Analysis of glycated haemoglobin was determined in the Lab of the University Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, Principal Investigator — University Complutense of Madrid